CLINICAL TRIAL: NCT01839955
Title: A Phase I Study of Erlotinib in Combination With Quinacrine in Patients With Advanced Non-Small-Cell Lung Cancer
Brief Title: Erlotinib Hydrochloride and Quinacrine Dihydrochloride in Stage IIIB-IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neelesh Sharma MD PhD (Other)
Responsible Party: Sponsor-Investigator, Neelesh Sharma MD PhD, Principal Investigator, Case Comprehensive Cancer Center
Organization: Case Comprehensive Cancer Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CASE8512; NCI-2013-00599 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-04-23; First posted 2013-04-25 (Estimated); Last update posted 2016-10-31 (Estimated); Status verified 2016-10

CONDITIONS: Recurrent Non-small Cell Lung Cancer; Stage IIIB Non-small Cell Lung Cancer; Stage IV Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Quinacrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Dose Escalation Group) (Experimental): Erlotinib hydrochloride and quinacrine dihydrochloride. The first three or six patients will be entered in this part of the study. Then this part will end.
  Interventions: Drug: erlotinib hydrochloride; Drug: quinacrine dihydrochloride - Escalation dose; Other: laboratory biomarker analysis; Other: pharmacological study
- Arm II (Extension Group) (Experimental): Erlotinib hydrochloride and quinacrine dihydrochloride. The next 12 patients will enter into the second part of this study.
  Interventions: Drug: erlotinib hydrochloride; Other: laboratory biomarker analysis; Other: pharmacological study; Drug: quinacrine dihydrochloride - Extension dose

INTERVENTIONS:
Drug: erlotinib hydrochloride — Dose Escalation Group:
  Begins day 1: given 150mg daily, orally
  Extension Group:
  Begins Day 1: 150mg daily, orally
  Other Names: CP-358,774; erlotinib; OSI-774
Drug: quinacrine dihydrochloride - Escalation dose — Begins Day 8: Loading dose (first cycle only) 50mg three times daily for 7 days followed by 21 days of 50mg maintenance dose. Level -1: Loading dose (50mg three times daily for 7 days), maintenance dose (50mg every other day for three weeks). Level 1 [starting dose]: Loading dose (50mg three times daily for 7 days), maintenance dose (50mg daily for three weeks). Level 2: Loading dose (100mg three times daily for 7 days), maintenance dose (100mg every other day for three weeks). Level 3: Loading dose (150mg three times daily for 7 days), maintenance dose (200mg every other day for three weeks). Level 4: Loading dose (200mg three times daily for 7 days), maintenance dose (400mg every other day for three weeks). Subsequent patient cohort(s) will be enrolled depending on the safety and tolerability of subjects
  Other Names: atabrine dihydrochloride; mepacrine dihydrochoride; SN 390
  Arms: Arm I (Dose Escalation Group)
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Drug: quinacrine dihydrochloride - Extension dose — Participants will be treated at recommended dose from expansion group to confirm tolerability and evaluate early response
  Other Names: atabrine dihydrochloride; mepacrine dihydrochoride; SN 390
  Arms: Arm II (Extension Group)

SUMMARY:
This phase I trial studies the side effects and best dose of quinacrine dihydrochloride when given together with erlotinib hydrochloride and to see how well it works in treating patients with stage IIIB-IV non-small cell lung cancer. Erlotinib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as quinacrine dihydrochloride, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving erlotinib hydrochloride together with quinacrine dihydrochloride may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety and tolerability of the combination of erlotinib (erlotinib hydrochloride) and quinacrine (quinacrine dihydrochloride) in patients with advanced non-small-cell lung cancer.

II. To determine the recommended Maximum Tolerated Dose (MTD) of the combination of erlotinib and quinacrine in patients with advanced non-small-cell lung cancer.

SECONDARY OBJECTIVES:

I. To describe the dose limiting toxicity of the erlotinib and quinacrine combination.

II. To determine the pharmacokinetic profile of the erlotinib and quinacrine combination.

III. To determine objective response rate (complete response [CR]+partial response [PR]) and clinical benefit rate (CR+PR+ stable disease [SD]) of the erlotinib and quinacrine combination.

IV. To estimate overall survival (OS)

OUTLINE: This is a phase I, dose escalation study of quinacrine dihydrochloride

Escalation Portion: Patients receive erlotinib hydrochloride orally (PO)daily on days 1-28 and quinacrine dihydrochloride PO thrice daily (TID) on days, 1-7 and PO daily from days 8-28.

After Maximum Tolerated Dose is established: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive erlotinib hydrochloride PO daily on days 1-28.

ARM II: Patients receive erlotinib hydrochloride PO and quinacrine dihydrochloride PO daily (TID) on days, 1-7 and PO daily from days 8-28.

In both arms, courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed incurable malignancy that is surgically unresectable locally advanced, recurrent, or metastatic (stage IIIB/IV) non-small cell lung cancer (NSCLC). Patients with adenocarcinoma, squamous cell carcinoma, large cell carcinoma and sarcomatoid carcinoma will be eligible.
* Patients must have received at least one platinum-containing regimen for the treatment of advanced or metastatic disease (except for EGFR-mutant patients). Prior maintenance therapy is allowed and will be considered as the same line of therapy when continued without discontinuation after initiation of a treatment regimen. NSCLC with documented EGFR mutation will be eligible after progression on an EGFR-TKI alone. NSCLC with other molecular targets, such as fusion gene involving the anaplastic lymphoma kinase (ALK) gene (such as echinoderm microtubule associated protein like 4 [EML4]-ALK) or ROS-1 will be eligible if they have progressed on targeted agents (ALK inhibitor) and chemotherapy or are not a candidate for chemotherapy. Adjuvant/neoadjuvant chemotherapy or chemoradiation is considered a line of therapy if < 12 months have elapsed between the last dose and the date of recurrence. Combined treatment with chemotherapy and radiation constitutes a single regimen.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Life expectancy of ≥ 12 weeks, in the opinion of and as documented by the investigator
* Hemoglobin ≥ 9.0 g/dl (transfusion and/or growth factor support allowed)
* Absolute neutrophil count (ANC) ≥ 1,500/mcL
* Platelet count ≥ 100 x 10^9 L
* Alkaline phosphatase < 2.5 X institutional upper limit of normal (in subjects with no liver metastasis and < 5.0 upper limit of normal [ULN] in subjects with liver metastasis)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) < 2.5 X institutional upper limit of normal (in subjects with no liver metastasis and < 5.0 ULN in subjects with liver metastasis)
* Serum creatinine ≤ 1.5 x ULN or creatinine clearance ≥ 50 mL/min
* Serum total bilirubin ≤ 1.5 x ULN OR total bilirubin ≤ 4.0 ULN with direct bilirubin ≤ 1.5 x ULN in patients with well documented Gilbert syndrome
* Patients who are receiving therapeutic anticoagulation with heparin are allowed to participate provided that no prior evidence of underlying abnormality exists in these parameters. Patients on warfarin are eligible provided they are on stable doses of warfarin and there is close monitoring of INR.
* Resolution of any toxic effects of prior therapy (including radiotherapy) according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.0, grade ≤ 1 (with the exception of alopecia and ≤ grade 2 neuropathy); subject must have recovered from significant surgery-related complications
* Women of childbearing potential must have a negative pregnancy test performed within 48 hours prior to the start of the study drug
* Women of child-bearing potential and men must agree to use adequate contraception (double barrier method of birth control or abstinence) prior to study entry, for the duration of study participation and for 90 days after completing the last investigational drug dose; should a woman become pregnant or suspect that she is pregnant while she or her partner is participating in this study, she should inform the treating physician immediately
* Subjects must have the ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients with previous anti-cancer chemotherapy, immunotherapy or investigational agents ≤ 3 weeks prior to the first day of study defined treatment. NSCLC patients with EGFR mutation can enroll within 7 days of discontinuing EGFR-TKI. Palliative radiation < 1 week before the start of treatment (lesions subjected to radiotherapy may not be used as target lesions). Patients who receive gamma knife radiosurgery for brain metastases within 1 week prior to treatment start.
* Patients with unknown status of EGFR mutation (only for patients with adenocarcinoma histology)
* Patients that have had major surgery ≤ 3 weeks or minor surgery (e.g. talc pleurodesis, excisional biopsy, etc) ≤ 1 week prior to the first day of study defined treatment.
* History of cardiac disease: congestive heart failure defined as class II to IV per New York Heart Association (NYHA) classification; active coronary artery disease (CAD); previously diagnosed bradycardia or other cardiac arrhythmia defined as ≥ grade 2 according to NCI-CTCAE (version 4.0), or uncontrolled hypertension; myocardial infarction occurred within 6 months prior to study entry (myocardial infarction occurred > 6 months prior to study entry is permitted)
* Patients with clinically unstable central nervous system (CNS) metastasis (to be enrolled in the study, subjects must have confirmation of stable disease by magnetic resonance imaging [MRI] or computed tomography [CT] scan within 4 weeks of the first day of study defined treatment and have CNS metastases well controlled by steroids, anti-epileptics or other symptom-relieving medications)
* Patients with significant gastrointestinal disorder that, in the opinion of the investigator, could interfere with absorption of quinacrine and/or erlotinib (eg, Crohn's disease, small or large bowel resection, malabsorption syndrome)
* Patients with any known contraindication to treatment with, including hypersensitivity to quinacrine or erlotinib
* Patients with active clinically serious infections defined as ≥ grade 2 according to NCI CTCAE, version 4.0
* Patients with substance abuse, medical, psychological or social conditions that may, in the opinion of the Investigator, interfere with the patient's participation in the study or evaluation of the study results
* Any other condition that is unstable or which could jeopardize the safety of the patient and his/her protocol compliance
* History of incurable malignancy other than NSCLC within the 5 years prior to start of treatment, with the exceptions of adequately treated intraepithelial carcinoma of the cervix uteri; prostate carcinoma with a prostate-specific antigen value <0.2 ng/mL; or basal or squamous-cell carcinoma of the skin.
* Pregnant or breastfeeding women and adults of reproductive potential not employing an effective method of birth control are excluded from this study because quinacrine is category N agent with the potential for teratogenic or abortifacient effects; these potential risks may also apply to other agents used in this study
* Patients with previously known infection with human immunodeficiency virus (HIV) or active viral hepatitis are ineligible because of the potential for pharmacokinetic interactions with quinacrine; (diagnostic testing for these infections will be done only if clinically indicated)
* Patients with known Glucose-6-phosphate deficiency, psoriasis, porphyria and psychosis (quinacrine may exacerbate the symptoms of these disorders)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-09; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of quinacrine dihydrochloride in combination of erlotinib hydrochloride determined by dose-limiting toxicities | 28 days
Progression Free Survival (PFS) | Date of randomization to the date of disease progression or the date of death, assessed up to 2 years
  Estimated by Kaplan-Meier method and the difference between two treatment arms will be evaluated by log-rank test.

SECONDARY OUTCOMES:
Pharmacokinetic parameters | after 2 months (2 cycles)
Objective tumor response rate (ORR) (complete response and partial response) evaluated by revised Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria | Up to 2 years
  Estimated based on the number of responses by excluding the dropouts who are not evaluable for response using a binomial distribution.
Disease stabilization rate (complete response, partial response and stable disease) | Up to 2 years
  The confidence intervals for them will be estimated using Wilson's method.
Baseline expression of intracellular inhibitor of the nuclear factor kappa B (IkappaB) or NFkappaB gene signature in determining survival or response | Baseline up to 2 years
Overall survival (OS) | Date of randomization to the date of death, assessed up to 2 years
  Estimated by Kaplan-Meier method and the difference between two treatment arms will be evaluated by log-rank test. Identified by Cox model or extended Cox model. Chi-square test or Fisher's exact test will be used to examine the difference of response rate between two treatment arms.

CONTACTS AND LOCATIONS:
Overall Officials: Neelesh Sharma, MD, PhD, Principal Investigator — University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- University Hospitals Cleveland Medical Center, Seidman Cancer Center, Case Comprehensive Cancer, Cleveland, Ohio, United States